CLINICAL TRIAL: NCT06945913
Title: The Effect Of Variable Intensity Swimming Exercise On Cardiovascular Parameters And Echocardiography In Women With Diastolic Dysfunction
Brief Title: Effect of Swimming Exercise on Diastolic Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Merve BOZ CİNCİ, Lecturer, Uşak University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UU-SBF-MBC-01
Record Dates: First submitted 2025-03-10; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Diastolic Dysfunction
Keywords: Diastolic Dysfunction; Exercise; High Intensity Interval Training; Moderate Intensity Continuous Training; Women Health
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: The study was conducted with three groups:
  The first group (n=20) performed high-intensity interval training (HIIT) swimming exercises.
  The second group (n=20) performed moderate-intensity continuous training (MICT) swimming exercises.
  The control group (n=20) did not engage in any exercise intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HIIT Group (Active Comparator): The first group (n=20) performed high-intensity interval training (HIIT) swimming exercises.
  Interventions: Behavioral: Exercise
- MICT Group (Sham Comparator): The second group (n=20) performed moderate-intensity continuous training (MICT) swimming exercises.
  Interventions: Behavioral: Exercise
- Non exercise Group (No Intervention): The control group (n=20) did not engage in any exercise intervention.

INTERVENTIONS:
Behavioral: Exercise — HIIT Group
  Arms: HIIT Group; MICT Group

SUMMARY:
The aim of the study was to determine the rehabilitative effects of 12-week variable intensity swimming exercises on the cardiovascular system in women with diastolic dysfunction. Studies on how variable intensity swimming exercises contribute to the course of the disease in sedentary women with cardiovascular problems are limited. Previous studies generally consisted of studies on the effects of exercise applications on the cardiovascular system in different branches and their effects were determined.

DETAILED DESCRIPTION:
Nowadays, combating diseases caused by sedentary lifestyle habits is among the fundamental challenges faced by humanity. With technological advancements, individuals spend most of their time in a sedentary manner, while also consuming fast-food products, which negatively affect overall health. Due to physical inactivity, obesity often develops, and in the long term, cardiovascular health is adversely impacted. As a result, physicians frequently prescribe regular exercise. To prevent the onset of such diseases, individuals engage in various sports activities. Walking, dancing, swimming, and strength training exercises are among the most preferred physical activities.

Swimming, which has become one of the most popular sports branches in Turkey compared to previous years, is gaining increasing popularity. The fact that swimming allows individuals to have an enjoyable time while exercising makes it a sought-after activity. Swimming is not only practiced professionally but is also a preferred sport among sedentary individuals aiming for a healthy lifestyle. Considering the sustainability of the learning process in this discipline, it should not be overlooked that swimming can positively contribute to instilling exercise habits in sedentary individuals.

Swimming exercises actively engage large muscle groups. Regular training of these muscle groups leads to cardiovascular adaptations that enhance exercise capacity, endurance, and skeletal muscle strength, while also preventing the development of coronary artery disease (CAD) and alleviating symptoms in individuals with pre-existing cardiovascular conditions. Swimming, which encompasses speed, strength, endurance, continuity, agility, flexibility, and aesthetic qualities, is one of the few sports disciplines that allow for the development of all these attributes over time. The improvement of physical fitness attributes is not only due to movement but also to resistance developed against water. This is because water is denser than air, requiring greater effort, thereby enhancing all physical fitness parameters in proportion to training intensity. Studies indicate that swimming exercises work the core, head, back, and abdominal muscles simultaneously, producing similar beneficial effects on the cardiovascular and skeletal systems. Moreover, swimming is among the few physical activities that ensure the harmonious development of the entire body with a significantly lower risk of injury compared to other sports disciplines. The buoyancy effect of water reduces the load on the joints, thereby minimizing musculoskeletal strain and injury risks. Given that joint disorders and related mobility limitations frequently occur due to sedentary habits in older age, swimming exercises play a crucial role in minimizing potential injuries.

To sustain vital functions, the body operates as an integrated system. All organs and tissues actively participate in these processes, ensuring continuity of life. Similarly, all motion-related activities in daily life are maintained through the extraordinary synchronization of the human body. Particularly in the case of physical activity, the load on key systems is significantly higher. For instance, while the musculoskeletal system largely assumes the responsibility for movement, the nervous system provides movement commands, and the circulatory system supplies the necessary oxygen and energy. The circulatory system, which serves as the locomotive to ensure continuity in these systems, bears crucial responsibility, especially during exercise. It delivers and transports oxygenated blood to all necessary points, a process facilitated by the superior anatomy of the heart. If the heart fails to pump blood, the entire body ceases to function. Furthermore, blood is essential for delivering the necessary nutrients to muscles during movement. The iron level in the human body significantly affects cardiovascular health, and both deficiencies and excesses can lead to severe complications . According to statistics from the Turkish Statistical Institute (TÜİK), circulation-related diseases ranked first in 2022, accounting for 35.4% of all cases. Among the 504,839 individuals included in the study, 178,501 died due to circulatory system diseases, 88,563 of whom were women.

Deterioration of heart health frequently leads to diastolic dysfunction, which is commonly associated with chronic hypertension, aging, particularly female gender, obesity, diabetes, chronic kidney disease, and cardiovascular diseases. High levels of LDL cholesterol and triglycerides in the blood play a significant role in the development of cardiovascular diseases. Studies have demonstrated that regular aerobic exercise, performed at controlled intensity levels, reduces triglycerides, total cholesterol, and LDL cholesterol while increasing HDL cholesterol, which benefits heart health.

Experimental studies have indicated that aging is associated with an increased risk of diastolic dysfunction in the heart. Aging is linked to numerous changes and adaptations in the cardiovascular system. While vascular and ventricular wall thickness increases, arterial compliance, endothelial function, and ventricular contractility decrease. Studies have reported that individuals who engage in regular exercise exhibit functional adaptations in heart performance, leading to a minimally enlarged and stronger heart. Consequently, due to the increased demand for blood during exercise, the heart's pumping capacity and cardiac output are enhanced. Research also indicates that physical activities with varying intensity levels improve well-being among adults while reducing the risk of cardiovascular diseases and cancer.

Although exercise is known for its many positive effects on the human body, individuals often lose interest over time. While exercise is expected to be an integral part of life, it gradually shifts away from becoming a routine. The primary reason for this decline is cited as lack of time. Historically, exercises recommended by medical experts for health improvement have involved continuous, moderate-intensity training over long periods, which can eventually lead to boredom or time constraints for individuals. One such exercise type is MICT (Moderate Intensity Continuous Training), characterized by continuous moderate-intensity workouts, typically performed at 50-60% intensity for durations ranging between 20-40 minutes. However, recent research suggests that short-duration, high-intensity interval training (HIIT) can also yield significant health benefits. HIIT, known as High-Intensity Interval Training, is increasingly recognized as a viable exercise option even for previously inactive individuals. HIIT is highly adaptable and can be implemented across various exercise domains. Due to its flexibility and efficiency, HIIT is frequently incorporated into exercise programs across different demographics. Given that many individuals struggle with time constraints, the shorter duration of HIIT sessions presents an opportunity for those with busy schedules to engage in regular exercise.

ELIGIBILITY:
Inclusion Criteria

Participants who met the following criteria were included in the study:

* No echocardiographic abnormalities detected except for stage 1 diastolic dysfunction based on examinations conducted in the cardiology outpatient clinic,
* Female gender,
* Aged between 40 and 60 years as of the study initiation date,
* No history of substance use, including smoking and alcohol,
* Willingness to participate by completing the informed consent form.

Exclusion Criteria

Participants who met at least one of the following conditions were excluded from the study:

* Refusal to sign the informed consent form,
* Failure to participate in at least one of the study measurements,
* Inability to meet the necessary criteria for training and measurements,
* Presence of illness or injury during training or measurements,
* Voluntary withdrawal from the study.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Heart Rate Measurement by Electrocardiography | 6 months
  Heart rate will be measured using a GE Healthcare MAC 2000 ECG device after 10 minutes of rest.
  Unit of Measure: Beats per minute (bpm)
P Wave Duration | 6 months
  The duration of the P wave will be measured using standard 12-lead ECG recordings.
  Unit of Measure: Milliseconds (ms)
PR Interval | 6 months
  The PR interval will be measured using standard 12-lead ECG recordings. Unit of Measure: Milliseconds (ms)
QRS Duration | 6 months
  The QRS duration will be measured using standard 12-lead ECG recordings. Unit of Measure: Milliseconds (ms)
QT Interval | 6 months
  The QT interval will be measured using standard 12-lead ECG recordings. Unit of Measure: Milliseconds (ms)
Corrected QT Interval (QTc) | 6 months
  The corrected QT interval (QTc) will be measured using standard 12-lead ECG recordings.
  Unit of Measure: Milliseconds (ms)

SECONDARY OUTCOMES:
Cardiac Cavity Dimensions by Echocardiography | 6 months
  Left ventricular internal diameter, left atrial size, and other cardiac cavity dimensions will be measured using Philips transthoracic echocardiography.
  Unit of Measure: Millimeters (mm)
Interventricular Septal Thickness | 6 months
  Measurements of interventricular septal thickness at end-diastole will be taken using echocardiography.
  Unit of Measure: Millimeters (mm)
Posterior Wall Thickness | 6 months
  Measurements of posterior wall thickness at end-diastole will be taken using echocardiography.
  Unit of Measure: Millimeters (mm)
Systolic Function - Ejection Fraction | 6 months
  Left ventricular systolic function will be evaluated using ejection fraction (EF) by the modified Simpson method.
  Unit of Measure: Percentage (%)
Diastolic Function - Early Diastolic Filling Velocity (E) | 6 months
  Early diastolic filling velocity will be measured using Doppler and tissue Doppler imaging.
  Unit of Measure: Centimeters per second (cm/s)
Diastolic Function - Late Diastolic Filling Velocity (A) | 6 months
  Late diastolic filling velocity will be measured using Doppler and tissue Doppler imaging.
  Unit of Measure: Centimeters per second (cm/s)
Diastolic Function - E/A Ratio | 6 months
  The ratio of early to late diastolic filling velocity (E/A) will be calculated. Unit of Measure: Unitless
Diastolic Function - Isovolumic Relaxation Time (IVRT) | 6 months
  Isovolumic relaxation time will be measured using Doppler and tissue Doppler imaging.
  Unit of Measure: Milliseconds (ms)
Diastolic Function - Deceleration Time (DT) | 6 months
  Deceleration time will be measured using Doppler and tissue Doppler imaging. Unit of Measure: Milliseconds (ms)
Diastolic Function - Early Myocardial Tissue Velocity (Em) | 6 months
  Early myocardial tissue velocity will be measured using tissue Doppler imaging. Unit of Measure: Centimeters per second (cm/s)
Diastolic Function - Late Myocardial Tissue Velocity (Am) | 6 months
  Late myocardial tissue velocity will be measured using tissue Doppler imaging. Unit of Measure: Centimeters per second (cm/s)
Diastolic Function - Em/Am Ratio | 6 months
  Description: The ratio of early to late myocardial tissue velocity (Em/Am) will be calculated.
  Unit of Measure: Unitless
Diastolic Function - E/Em Ratio | 6 months
  The ratio of early diastolic filling velocity to early myocardial tissue velocity (E/Em) will be calculated.
  Unit of Measure: Unitless

CONTACTS AND LOCATIONS:
Locations (1):
- Uşak U, Uşak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No